CLINICAL TRIAL: NCT01694888
Title: Midwifery Students' Performance Before and After Teaching Fundamentals of Documentation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, nazila zarghi, faculty member, Mashhad University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Documentation Skill
Record Dates: First submitted 2012-09-17; First posted 2012-09-27 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2011-04

CONDITIONS: Documentation Skill
Keywords: Students practice, Lecture; Nursing records; Nursing education; Midwifery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- midwifery students (Experimental): all midwifery students studying at last term (except one who was absent) (27) in Mashhad school of nursing and midwifery in April 2011
  Interventions: Other: lecture

INTERVENTIONS:
Other: lecture — Teaching documentation skill using lecture method

SUMMARY:
Midwives are responsible for documenting and keeping care facts in midwifery departments. Inaccurate documentation or even minute error in reporting may lead to burdensome responsibility for midwives. This study has been conducted aimed to compare midwifery students' performance before and after teaching fundamentals of documentation. In this quasi-experimental study, 28 midwifery students were participated. Data were collected by a questionnaire including a. demographic data and b. Scenarios (1) and (2) of an imaginary patient with physician order and a checklist contain 11 elements of documentation

ELIGIBILITY:
Inclusion Criteria:

* midwifery students studying at mashhad school of nursing and midwifery

Exclusion Criteria:

* any other discipline

Ages: 21 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
compare midwifery students' performance before and after teaching fundamentals of documentation using lecture method | up to one month